CLINICAL TRIAL: NCT05471544
Title: Effectiveness, Feasibility and Acceptability of Seasonal Malaria Chemoprevention in Aweil South County in Northern Bahr Eel Ghazal, South Sudan: A Type 2 Hybrid Effectiveness-implementation Study Using a Convergent Mixed-methods Approach
Brief Title: Effectiveness, Feasibility and Acceptability of Seasonal Malaria Chemoprevention in Aweil South County in South Sudan
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Malaria Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMCSSPHASE1
Record Dates: First submitted 2022-07-15; First posted 2022-07-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-10

CONDITIONS: Malaria
Keywords: seasonal-malaria-chemoprevention
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sulfadoxine-Pyrimethamine + Amodiaquine (SPAQ) (Experimental): Children aged 3-59 months will receive SPAQ in the intervention arm
  Interventions: Drug: Sulfadoxine pyrimethamine; Drug: Amodiaquine
- Control (No Intervention): Children aged 3-59 months will not receive SPAQ in the control arm

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine — Sulphadoxine is a slowly eliminated sulphonamide. It is used in a fixed dose combination of 20 parts sulphadoxine with 1 part pyrimethamine given orally or intramuscularly.
  The medicine is no longer recommended for the treatment of malaria. However, it is being used for Intermittent Preventive Treatment during pregnancy (IPTp) and as a co-packaged combination with amodiaquine for seasonal malaria chemoprevention.
  Sulphadoxine is readily absorbed from the GIT. It is widely distributed in body tissues and fluids and crosses the placenta into foetal circulation. It is also readily detectable in breast milk. It is excreted predominantly as the unchanged drug.
  Other Names: SP
  Arms: Sulfadoxine-Pyrimethamine + Amodiaquine (SPAQ)
Drug: Amodiaquine — Amodiaquine is a Mannich base 4 amino-quinoline that interferes with parasite haem detoxification. It is more effective than chloroquine in both chloroquine sensitive and resistant P. falciparum infections. However, there is cross-resistance between chloroquine and amodiaquine.
  It is readily absorbed in the GIT and rapidly converted in the liver to the active metabolite, desethylamodiaquine. Desethylamodiaquine is responsible for all the antimalarial effect.
  Other Names: AQ
  Arms: Sulfadoxine-Pyrimethamine + Amodiaquine (SPAQ)

SUMMARY:
This study aims to explore whether SMC is an effective intervention in the context of Northen Bahr el Gazal state, South Sudan. It also aims to assess the protective efficacy of the antimalarials used in SMC in the target population and investigate levels of parasite resistance in the study counties. If successful, this trial should provide the evidence for SMC to be included in malaria programming and policy in South Sudan.

A Type II hybrid effectiveness-implementation study design will be used to evaluate the effects of a clinical intervention on relevant outcomes whilst collecting information on implementation. It is designed to determine feasibility and effectiveness of an innovative intervention, as well as the protective efficacy of the antimalarial drugs used. The study consists of five components: 1) A series of cross-sectional surveys establishing confirmed malaria cases in children; 2) A prospective cohort study to determine the protective efficacy of SPAQ (if SPAQ provides 28 days of protection from infection) and whether drug concentrations and/or resistance influence the duration of protection; 3) A resistance markers study in children 3-59 months in the research county; 4) Modelling the protective effect of SPAQ in South Sudan to determine where SMC could be a suitable malaria prevention strategy in other areas of the country, and 5) A process evaluation to understand feasibility and acceptability of the SMC intervention in South Sudan.

DETAILED DESCRIPTION:
This is an implementation research study, using a Type II hybrid effectiveness-implementation study design, to evaluate the effects of a clinical intervention on relevant outcomes whilst collecting information on implementation.

The study uses pragmatic implementation research with the objective of contributing to the development of practical recommendations for health policy, practice and potential scale up. It is designed as an implementation study to determine effectiveness and protective efficacy to gather evidence of its potential impact on health outcomes. Five monthly cycles of SMC will be implemented between June and October 2022 in one county, Aweil South, in Northern Bahr el Gazal state.

The study will comprise the following six components :

1. Two cross-sectional surveys at the height of the malaria season to explore impact on malaria incidence
2. End-of-round survey
3. Prospective protective efficacy cohort study to determine if SPAQ provides 28 days of protection from infection and whether drug concentrations and/or resistance influence the duration of protection
4. Resistance markers study in children 3-59 months in the two research counties plus the two standard intervention counties to measure changes in resistance marker prevalence over time (pre and post within the same year and between years)

ELIGIBILITY:
Inclusion Criteria:

* Being resident in the project area
* Afebrile with no other malaria associated symptoms in the past 48 hours or at time of recruitment
* Consent to participate in the study obtained
* Can comply with 3 day DOT of standard SPAQ regimen (day 0-2)
* Willingness and ability of the childs guardians to comply with the study protocol for the duration of the study including all dry blood spot and slide collections

Exclusion Criteria:

* Symptoms of malaria (tympanic fever ≥ 37.5 °C or history of fever in past 48 hours)
* Known allergy to medicine provided
* Receiving a sulfa-based medication for treatment or prophylaxis, including co-trimoxazole (trimethoprim-sulfamethoxazole).
* Individuals receiving azithromycin due to the antimalarial activity of azithromycin.
* Severe malnutrition according to WHO guidelines
* Recruited in cross sectional surveys or any other SMC studies.
* Children with HIV
* Previous treatment with Amodiaquine in the past 28 days (treatment with ASAQ or SPAQ)

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3575 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Malaria incidence in study population in intervention county and eligible children in one control county | Five months
  Number of malaria cases in the intervention population and eligible children in one control county over the study period as reported through care givers in cross-sectional surveys at baseline, mid-intervention and endline
Chemoprevention failure as defined by positive parasites in malaria slides after day 7 or positive qPCR in dried blood spot (DBS) on day 28 | One month
  Malaria slides and dry blood spots (DBS) taken at days 0,7, 28 will be analysed with qPCR methodology to detect low level submicroscopic parasitemia in children treated with SPAQ
Prevalence of antimalarial resistance markers (dhfr, dhps, Pfcrt, pfmdr1) among chemoprevention failures as defined in outcome 2 | One month
  All Dried blood spots (DBS) will be analysed for malaria mutation genotypes (dhfr, dhps, Pfcrt, pfmdr1) on baseline and endline and additionally on day 7, day 28, or if participant slide is positive for parasites on day 7 or an infection is reported through care givers in cross-sectional survey.
Drug concentrations of Sulfadoxine-pyrimethamine and amodiaquine among chemoprevention failures (as defined in outcome 1) | One month
  Drug concentrations will be analyzed for all samples on baseline, day 7 and day 28 and will be linked to chemoprevention failure cases as defined in outcome 2 or a malaria infection is reported through care givers in cross sectional survey.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ismail Julla, Principal Investigator — Ministry of Health, South Sudan
Locations (1):
- Aweil South, Aweil, Northern Bahr El Gazal, South Sudan

IPD SHARING:
Plan to Share IPD: No
As this data is sensitive we propose not to share it.